CLINICAL TRIAL: NCT05306652
Title: Exercise in Extended Oncogene Addicted Lung Cancer in Active Treatment: a Randomized Controlled Trial
Brief Title: Exercise in Extended Oncogene Addicted Lung Cancer in Active Treatment
Acronym: EXcellenT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AUSL Romagna Rimini (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EXcellenT
Record Dates: First submitted 2022-02-22; First posted 2022-04-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Oncogene addiction; physical activity; personalized
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Oncogene Addiction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Home based supervised physical exercise (Experimental): patients will have a home-based physical activity prescription
  Interventions: Other: Supervised physical activity
- B- Unsupervised physical exercise (Active Comparator): patients will receive a physical activity counselling, without a real prescription and supervision
  Interventions: Other: Unsupervised physical activity

INTERVENTIONS:
Other: Supervised physical activity — patients will have a home-based physical activity prescription, defined on the functional endurance and strength tests and they will be supervised for 3 months. Once monthly they will be examined by the oncologist (visit and questionnaires) and at weeks 4, 6, 8, 10 and 12 at the sport medicine center where the three tests will be repeated. Home-based activity will be monitored daily through a specific application. Endurance improvement is defined as an increase in walking speed; strength improvement is defined as an increase of the number of repetitions
  Arms: A - Home based supervised physical exercise
Other: Unsupervised physical activity — patients will receive a physical activity counselling, without a real prescription and supervision, and the three test will be repeated once a month for three months at the local sport medicine center and at the oncology center (visit and questionnaires). Counselling will include general informations on physical exercise
  Arms: B- Unsupervised physical exercise

SUMMARY:
This is an interventional, non-pharmacologic, randomized controlled study evaluating the impact on quality of life of a personalized exercise program in oncogene addicted lung cancer patients undergoing active treatment. Patients will be randomized 1:1 in two arms: arm A (interventional) and arm B (control). The program of physical activity will be established after a test done at the local clinical center and based on easy exercises already studied in other diseases (e.g. coronary syndrome or organ transplant). A smartphone application will allow patients to register their daily physical activity and to easily recover data on strength and endurance. Patients in Arm A will have a home-based physical activity prescription and will be supervised at weeks: 4, 6, 8, 10, 12 by the oncologist and an exercise expert of the local sport center through three exercises (body composition test, endurance test and strength test) and questionnaires. Home-based activity will be monitored daily though a specific application (provided by Technogym). Patients in Arm B will receive an exercise counselling without a subsequent supervision. The three tests and questionnaires will be repeated once a month for three months at the local sport center and oncology center. Counselling will include general information on exercise. Patients will undergo blood sampling at baseline, week 4 and week 12 in order to evaluate changes in their immunological state (lymphocyte populations and cytokines).

DETAILED DESCRIPTION:
This is an interventional, non pharmacological, randomized controlled trial evaluating the impact on quality of life of a personalized exercise program in oncogene addicted lung cancer patients undergoing active treatment.

At Baseline every patient will receive three tests at the Division of Sport Medicine of Azienda Unità Sanitaria Locale (AUSL) of Romagna (Ravenna)

1. Body composition Analysis: Height, Weight, Bioimpedentiometry (resistance and reactance), Volume of Oxygen (VO2) max.
2. Endurance test: 1 Km treadmill test.
3. Strength test: Repetition of three different exercises (Chest press - upper limbs; Leg press - lower limbs; Lat pull down or Lat Machine or Upper Back).

After the three tests have been performed patients will be evaluated for eligibility and randomized into two arms: Arm A (interventional) and Arm B (control).

The program will be guided (prescribed and supervised) by an oncologist and a sport medicine doctor.

Arm A (interventional): patients will have a home-based physical activity prescription, defined on the functional endurance and strength tests and they will be supervised for 3 months. Once monthly they will be examined by the oncologist (visit and questionnaires) and at weeks 4, 6, 8, 10 and 12 at the sport medicine center where the three tests will be repeated. Home-based activity will be monitored daily through a specific application (provided by Technogym). Endurance improvement is defined as an increase in walking speed; strength improvement is defined as an increase of the number of repetitions.

Arm B (control): patients will receive a physical activity counselling, without a real prescription and supervision, and the three test will be repeated once a month for three months at the local sport medicine center and at the oncology center (visit and questionnaires). Counselling will include general informations on physical exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Willingness to provide written informed consent.
3. Life expectancy >12 weeks.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
5. Body massa index > 18.
6. Oncogene-addicted (EGFR, ALK, ROS1, RET, BRAF) stage IV or III b not suitable for local treatment receiving first- or second-line systemic treatment (palliative radiotherapy and prior chemotherapy allowed). Patients undergoing treatment in clinical trials are excluded.

Exclusion Criteria:

1. Inability to walk.
2. Immobility for more than 3 days before study enrollment.
3. Previously untreated (non-irradiated or non-resected) symptomatic brain metastases.
4. Severe cardiac impairment (e.g. cardiac insufficiency New York Heart Association (NYHA) > III, myocardial infarction within the last three months, severe cardiac arrhythmias, high grade aortic stenosis).
5. Severe respiratory failure.
6. Uncontrolled pain.
7. Bone metastasis inducing increased risk of pathological fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Impact of personalized prescription of physical exercises on quality of life assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) | 12 weeks
  To evaluate the impact of a personalized prescription of physical exercises monitored through a special smartphone application on quality of life assessed with the Italian version of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30)
Impact of personalized prescription of physical exercises on quality of life assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire for lung cancer (QLQ-LC29) | 12 weeks
  To evaluate the impact of a personalized prescription of physical exercises monitored through a special smartphone application on quality of life assessed with the Italian version of the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire for lung cancer (QLQ-LC29)
Impact of personalized prescription of physical exercises on quality of life assessed by the Beck Depression Inventory II (BDI-II) | 12 weeks
  To evaluate the impact of a personalized prescription of physical exercises monitored through a special smartphone application on quality of life assessed with the Italian version of Beck Depression Inventory II (BDI-II)

SECONDARY OUTCOMES:
Adherence to prescription | 12 weeks
  To evaluate the adherence to the step-counter and the strength training prescription monitored through a specific smartphone application. the number of weeks (at least 9 out of 12 weeks) a subject follows the personalized activity prescription will be measured
change of functional capacity | 12 weeks
  Functional capacity will be measured through the 1 Km treadmill test (at baseline; at week 4, week 8 and at week 12): arm A versus arm B. For those in the experimental arm, as the individual progresses with the exercise plan, the exercise dosage will be modulated to facilitate improvements.
change of muscle strength | 12 weeks
  Muscle strength will be measured through the maximum repetition tests (at baseline; at week 4, week 8 and at week 12): arm A versus arm B. For those in the experimental arm, as the individual progresses with the exercise plan, the exercise dosage will be modulated to facilitate improvements.
tolerance to treatment | 12 weeks
  Monitoring the frequency, duration, and severity of adverse events (AEs), through physical examinations, changes in vital signs and through clinical laboratory blood.
Overall survival (OS) | 24 months
  Overall survival (OS), defined as the time from randomization to death from any cause.
Patient's satisfaction assessed by dedicated questionnaire | 12 weeks
  Patient's satisfaction of an App-based system to guide and monitor home-based physical activity is assessed by dedicated questionnaire addressing specific issues
impact of personalized exercise on immunity state | 12 weeks
  T Lymphocytes modulation during physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Bennati, Principal Investigator — AUSL Romagna
Locations (1):
- S.Maria delle Croci Hospital, Oncology Unit, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No